CLINICAL TRIAL: NCT00162253
Title: Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study of BMS-587101 in Patients With Moderate to Severe Psoriasis
Brief Title: Study of BMS-587101 in Patients With Moderate to Severe Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM117-005
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2007-09

CONDITIONS: Psoriasis, Moderate to Severe
MeSH Terms: conditions — Psoriasis | interventions — 5-(9-(4-cyanophenyl)-3-(3,5-dichlorophenyl)-1-methyl-2,4-dioxo-1,3,7-triazaspiro(4,4)non-7-ylmethyl)-3-thiophenecarboxylic acid

INTERVENTIONS:
Drug: BMS 587101

SUMMARY:
The purpose of this clinical research study is to learn if BMS-587101 is effective on the treatment of Moderate to Severe Psoriasis. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria: Otherwise healthy individuals with a diagnosis of plaque-type psoriasis at least 6 months prior to screening (subjects with concurrent psoriatic arthritis may be enrolled).

Men and Women Not of Child Bearing Potential (i.e. women who are postmenopausal or surgically sterile), women ages 18 to 75.

-

Exclusion Criteria: Women of Child Bearing Potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study.

Known or suspected infection, including infection with human immunodeficiency virus (HIV), hepatitis B or C viruses. Any recent infections requiring antibiotic treatment that completed within 4 weeks of enrollment.

Any known malignancy or history of malignancy within 5 years prior to enrollment, with the exception of basal cell or squamous cell carcinoma of the skin that has been excised with no evidence of recurrence (squamous cell carcinoma of other locations is exclusionary).

Any history of Guillane-Barre syndrome. History of keloid formation.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-04; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To estimate the clinical response in terms of the percent of subjects achieving PASI_50 in each treatment arm, and to determine whether there was a difference in PASI_50 between each BMS-587101 treatment arm and placebo

SECONDARY OUTCOMES:
To estimate the proportion of patients achieving a PASI 75 response in each treatment arm.
To estimate the percent change (or reduction) in PASI score at 12 weeks of treatment in each treatment arm.
To estimate the proportion of patients achieving a PGA score of clear to minimal in each treatment arm.
To estimate the percent change from baseline in epidermal thickness of psoriatic lesion.
To evaluate the safety and tolerability of BMS-587101 in patients with psoriasis.
To evaluate the single- and multiple-dose pharmacokinetics of BMS-587101

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Local Institution, Phoenix, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, San Diego, California
  - Local Institution, Miami Beach, Florida
  - Local Institution, Pinellas Park, Florida
  - Local Institution, Boise, Idaho
  - Local Institution, Fridley, Minnesota
  - Local Institution, St Louis, Missouri
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, New York, New York
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Columbus, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Greer, South Carolina
  - Local Institution, Dallas, Texas